CLINICAL TRIAL: NCT03115190
Title: A Prospective Cohort Study to Improve the Accuracy of Referrals of Patients With Chest Pain to the Emergency Department: to Decrease the Delay in Acute Coronary Syndrome Patients and Rule Out Non-cardiac Chest Pain Patients (URGENT)
Brief Title: Improving the Referral of Patients With Chest Pain
Acronym: Urgent
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Philips Minicare has been taken off the market due to financial company issues that have nothing to do with the safety of the Minicare or the URGENT trial.
Sponsor: VieCuri Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Rahel2017Urgent
Record Dates: First submitted 2017-04-11; First posted 2017-04-14 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; Chest Pain
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- General practitioner diagnosis with Heart score (Other): Patients with chest pain who are reviewed by the general practitioner (GP) at the GP cooperation will be evaluated with the Heart score to support the GP with the diagnosis.
  Interventions: Diagnostic Test: General Practitioner diagnosis with Heart score
- Triage Nurse education (No Intervention): The general practitioner cooperation employs nurses for (telephone) triage. They are aided by a computer based triage system, the Netherlands triage system (NTS), a 6-level urgency triage system. With this study we aim to educate the nurses in the signs and symptoms of chest pain patients. The training program will aim to educate the triage nurses in acute coronary syndrome, including pathophysiology, symptoms and risk factors. The NTS will be incorporated within the training. The triage nurses will receive a training session by Cardiologists with information about acute coronary syndrome, the symptoms and the risks.
- Baseline registry as comparison (No Intervention): All patients referred to the emergency department (ED) with suspected acute coronary syndrome (ACS) will be evaluated. They will receive a questionnaire to evaluate the accuracy of referral and the delays of ACS patients. This will be compared to the registry at baseline. Some patients will either have not contacted the general practitioner cooperation (GPC) at all, or will have been referred to the ED directly through the GPC nurse triage.
  The 30 day, 6 months and one year follow-up of all patients will be via medical records, or in case of no or not enough information, by telephone.

INTERVENTIONS:
Diagnostic Test: General Practitioner diagnosis with Heart score — All patients seen by the general practitioner (GP) at the GP cooperation and agreeing to participation will be evaluated with the Heart score. This is a score including history, electrocardiogram, age, risk factors and troponin to assess whether a patient is at high risk for acute coronary syndrome. The troponins asked for in the Heart score are at arrival of the patient, not regarding the time of onset of chest pain. We shall use point of care (POC) troponin, thereby modifying the Heart score. The GP must realize that the POC troponin is not reliable on its own with one test. If the Heart score is low, it is acceptable and safe to not refer the patient, it is however not safe to refer the patient solely on negative troponin result.
  Arms: General practitioner diagnosis with Heart score

SUMMARY:
Rationale: This study aims to aid the general practitioner (GP) in the diagnostic dilemma of chest pain patients. Patients with acute coronary syndrome (ACS) should be referred to the hospital promptly, though referring all patients with chest pain is not feasible, as up to 80% of the patients with chest pain in the primary care do not have ACS.

Objective: The primary objective is to refer patients who contact the out-of-hours GP cooperation (GPC) with suspicion of ACS more accurately with a hypothesized reduction of 10% in unnecessary referrals.

Study design: This study is a prospective, observational, prevalence-based cohort study within the standard care of ACS patients.

Study population: All patients with chest pain, or other complaints suspect of ACS, will be included in which the GP at the GPC is in need of further diagnostics to come to a decision of referral. The follow-up will be a registry of all patients with suspected ACS referred to the emergency department (ED). Patients with typical complaints of ACS, and thus a high suspicion, will be excluded and referred promptly.

Intervention: Triage nurses working at the GPC will receive specific ACS training. Patients who arrive at the GPC with non-typical chest pain, will be screened for enrolment within the study. The GP evaluates patients using the Heart score, this includes electrocardiogram recording and point of care (POC) troponin testing. With the Heart score the GP can make an informed decision to refer the patient to the ED.

To evaluate the intervention a registry of all patients referred to the ED with suspected ACS will be compared to a baseline registry performed from the 1st of September 2015 until the 1st of March 2016. Patients not referred to the ED, will have a (standard) high-sensitivity troponin and a POC troponin as follow-up at least four hours (up to 24 hours) after first measurement.

The burden and risks associated with participation, benefit and group relatedness: Patients enrolled within this study will receive a finger stick blood test and electrocardiogram recording at the GPC and a finger stick blood test and a venous blood test at least four hours after first troponin measurement. We may follow-up by telephone if we can not obtain the required information from medical records. We expect no adverse events and there are no expected risks associated with this protocol. We expect patients with ACS to be referred more accurately and more promptly to the ED and thus lowering risks.

ELIGIBILITY:
Inclusion Criteria:

All patients with chest pain or other complaints suspect of acute coronary syndrome (ACS) can be included in which the general practitioner is in need of further diagnostics to come to a decision of referral.

All patients referred to the emergency department (ED) with suspected ACS will be included to evaluate the appropriateness of referral.

Exclusion Criteria:

* Patients younger than 18 years
* Patients in which a typical history and/or physical examination requires immediate referral; high suspicion of ACS
* Patients in which an acute non-coronary diagnosis is suspected, e.g. pulmonary embolism, thoracic aortic dissection etc.

The baseline of patients seen at the ED will not exclude any patients referred with suspected ACS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Suspected diagnosis | 30 days
  The primary outcome measure is a more accurate referral of patients with suspected acute coronary syndrome (ACS) to the cardiac emergency department and thus the concordance of suspected ACS and the actual diagnosis. The endpoint will be compared to the baseline registry that has been executed from 1st of September 2015 until 1st of March 2016.

SECONDARY OUTCOMES:
Major adverse cardiovascular events | 30 days, 6 months and 1 year
  Combination endpoint of: mortality and any ischemic event (ST-elevated myocardial infarction, non-ST-elevated myocardial infarction, (Unstable)Angina Pectoris, Percutaneous Coronary Intervention, Coronary Artery Bypass Grafting, Resuscitation)

CONTACTS AND LOCATIONS:
Locations (1):
- VieCuri Medical Center, Venlo, Netherlands

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to other researchers to secure privacy in study patients.

REFERENCES:
- [Background] Verdon F, Herzig L, Burnand B, Bischoff T, Pecoud A, Junod M, Muhlemann N, Favrat B; GMIRG. Chest pain in daily practice: occurrence, causes and management. Swiss Med Wkly. 2008 Jun 14;138(23-24):340-7. doi: 10.4414/smw.2008.12123. PMID 18561039
- [Background] Task Force on the management of ST-segment elevation acute myocardial infarction of the European Society of Cardiology (ESC); Steg PG, James SK, Atar D, Badano LP, Blomstrom-Lundqvist C, Borger MA, Di Mario C, Dickstein K, Ducrocq G, Fernandez-Aviles F, Gershlick AH, Giannuzzi P, Halvorsen S, Huber K, Juni P, Kastrati A, Knuuti J, Lenzen MJ, Mahaffey KW, Valgimigli M, van 't Hof A, Widimsky P, Zahger D. ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation. Eur Heart J. 2012 Oct;33(20):2569-619. doi: 10.1093/eurheartj/ehs215. Epub 2012 Aug 24. No abstract available. PMID 22922416
- [Background] Bosner S, Becker A, Haasenritter J, Abu Hani M, Keller H, Sonnichsen AC, Karatolios K, Schaefer JR, Seitz G, Baum E, Donner-Banzhoff N. Chest pain in primary care: epidemiology and pre-work-up probabilities. Eur J Gen Pract. 2009;15(3):141-6. doi: 10.3109/13814780903329528. PMID 19883149
- [Background] Ruddox V, Mathisen M, Otterstad JE. Prevalence and prognosis of non-specific chest pain among patients hospitalized for suspected acute coronary syndrome - a systematic literature search. BMC Med. 2012 Jun 12;10:58. doi: 10.1186/1741-7015-10-58. PMID 22691301
- [Background] Webster R, Norman P, Goodacre S, Thompson A. The prevalence and correlates of psychological outcomes in patients with acute non-cardiac chest pain: a systematic review. Emerg Med J. 2012 Apr;29(4):267-73. doi: 10.1136/emermed-2011-200526. Epub 2011 Oct 27. PMID 22034535
- [Background] Weinstock MB, Weingart S, Orth F, VanFossen D, Kaide C, Anderson J, Newman DH. Risk for Clinically Relevant Adverse Cardiac Events in Patients With Chest Pain at Hospital Admission. JAMA Intern Med. 2015 Jul;175(7):1207-12. doi: 10.1001/jamainternmed.2015.1674. PMID 25985100
- [Background] Knockaert DC, Buntinx F, Stoens N, Bruyninckx R, Delooz H. Chest pain in the emergency department: the broad spectrum of causes. Eur J Emerg Med. 2002 Mar;9(1):25-30. doi: 10.1097/00063110-200203000-00007. PMID 11989492
- [Background] Huibers L, Giesen P, Smits M, Mokkink H, Grol R, Wensing M. Nurse telephone triage in Dutch out-of-hours primary care: the relation between history taking and urgency estimation. Eur J Emerg Med. 2012 Oct;19(5):309-15. doi: 10.1097/MEJ.0b013e32834d3e67. PMID 22008589
- [Background] Nilsson S, Ortoft K, Molstad S. The accuracy of general practitioners' clinical assessment of chest pain patients. Eur J Gen Pract. 2008;14(2):50-5. doi: 10.1080/13814780802342622. PMID 18720273
- [Background] Wilcox HM, Vickery AW, Emery JD. Cardiac troponin testing for diagnosis of acute coronary syndromes in primary care. Med J Aust. 2015 Oct 19;203(8):336. doi: 10.5694/mja14.01154. PMID 26465699
- [Background] Backus BE, Six AJ, Kelder JC, Mast TP, van den Akker F, Mast EG, Monnink SH, van Tooren RM, Doevendans PA. Chest pain in the emergency room: a multicenter validation of the HEART Score. Crit Pathw Cardiol. 2010 Sep;9(3):164-9. doi: 10.1097/HPC.0b013e3181ec36d8. PMID 20802272
- [Background] Leite L, Baptista R, Leitao J, Cochicho J, Breda F, Elvas L, Fonseca I, Carvalho A, Costa JN. Chest pain in the emergency department: risk stratification with Manchester triage system and HEART score. BMC Cardiovasc Disord. 2015 Jun 11;15:48. doi: 10.1186/s12872-015-0049-6. PMID 26062607
- [Background] Ishak M, Ali D, Fokkert MJ, Slingerland RJ, Tolsma RT, Badings E, van der Sluis A, van Eenennaam F, Mosterd A, Ten Berg JM, van 't Hof AW. Fast assessment and management of chest pain patients without ST-elevation in the pre-hospital gateway (FamouS Triage): ruling out a myocardial infarction at home with the modified HEART score. Eur Heart J Acute Cardiovasc Care. 2018 Mar;7(2):102-110. doi: 10.1177/2048872616687116. Epub 2017 Jan 13. PMID 28084079